CLINICAL TRIAL: NCT02692573
Title: Prone or Supine Effect of Immediate Positioning After Scheduled Caesarean Delivery on Respiratory Outcomes in Full Term Infants
Brief Title: Prone or Supine Effect After Caesarean Delivery on Respiratory Outcomes in Full Term Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Montefiore Medical Center (Other)
Responsible Party: Principal Investigator, Thomas Havranek, Attending Neonatologist, Associate Professor of Pediatrics, Montefiore Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2015-5470
Record Dates: First submitted 2016-02-16; First posted 2016-02-26 (Estimated); Last update posted 2019-02-05 (Actual); Status verified 2019-02

CONDITIONS: Prone vs Supine Effects on Respiratory Outcomes
MeSH Terms: interventions — Patient Positioning

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- prone (Experimental): Prone positioned after delivery
  Interventions: Other: positioning
- supine (Active Comparator): Supine positioned after delivery
  Interventions: Other: positioning

INTERVENTIONS:
Other: positioning — prone positioning for the initial 5 minutes of life
  Arms: prone
Other: positioning — supine positioning for the initial 5 minutes of life
  Arms: supine

SUMMARY:
Investigators will compare 500 full term babies delivered by SCD randomized into two groups, prone or supine position. Investigators will use a Panda warmer with built in Nellcor pulse oximeter. Each infant will have heart rate (HR), oxygen saturation via pulse oximetry, respiratory rate and respiratory effort documented every 1 minute for the first 5 minutes of life; beyond the initial 5minutes of life, monitoring as well as infant's management will be done as per current Weiler hospital protocols. The intervention group will be placed in prone position for first five minutes immediately after birth, and then changed to supine position. The control group will be placed supine from birth. Investigators will check for the incidence and severity of RD, supplemental oxygen need and duration, positive pressure ventilation (PPV) need and duration or other use of respiratory support (intubation). Additionally, investigators will record the number of infants requiring admission to the NICU in each group, days of ventilatory support as well as the length of hospitalization.

DETAILED DESCRIPTION:
1. Consent obtained prior to actual operative delivery and anesthesia
2. Prior to start of surgery an opaque envelope with random selection of post delivery position, supine or prone, is opened
3. Pediatric team confirms with Obstetrician and delivery team the position in which the infant will be given to pediatrics
4. Pediatric team member accepting the infant stays by the operating room table to observe the delivery At actual delivery, the Panda radiant warmer Apgar clock will be started by a Pediatric team member positioned at the warmer when the baby is delivered. Vitals signs of HR, color and oxygen saturations will be recorded each minute for first five minutes. Respiratory effort will be noted. The Apgar clock is available to document the timing of the minute intervals heart rate and oxygen saturations on the preprinted grid of the survey data sheet.

6. When a Group A (supine) infant's transfer is made to Pediatrics, the infant will be kept in the supine position in transit to warmer and on warmer until first towel drying completed, 30 - 60 seconds, consistent with NRP protocol. Pulse oximetry and temperature probe will be placed. Vitals signs of HR, color and oxygen saturations will be recorded each minute for first five minutes. Respiratory effort will be noted.

When a Group B (start in prone position) the obstetrician places the baby in prone position, clamps and cuts cord. The baby is given to Pediatrics in the prone position. The infant will be kept in the prone position in transit to warmer and on warmer for first towel drying completed. Pulse oximetry and temperature probe will be placed. Vitals signs of HR, RR and oxygen saturations will be recorded each minute for first five minutes. Respiratory effort will be documented.

7. As toweling is changed the baby in prone position continues as such until five minutes pass. After five minutes the baby is turned to supine position as per standard NRP protocol.

8. Decision to initiate positive pressure ventilation and /or oxygen supplementation will be guided by published NRP 2010 lower saturation targets (1 min <60%, 2 min <65%, 3 min <70%, 4 min <75%, 5 min <80%) and/or by grunting, retractions ; discontinuation by high saturation targets (1min >65%, 2 min >70%, 3min >>75%, 4 min >80%, 5 min >85%) and resolution of respiratory distress. Positive pressure ventilation will be delivered via Neopuff device in supine position (both groups); CPAP 5cm 21% initially, then the amount of oxygen will be titrated to meet oxygen saturation target for given minute of life.

9. After no more than 30 minutes, Primary Assignment for admission to the NBN vs. NICU is made by a trained member of the study who was not in the operating room at the beginning of the delivery when the initial positioning of the infant was revealed. This is possible with 24 hour coverage from attendings, fellows, and mid-level practioners. Determination is based on Weiler NICU admission protocols.

10. If infant is to go to NBN then STS and breastfeeding protocols will be followed.

11. Infants developing respiratory distress in the NBN will be transferred to the NICU for further evaluation and care 12. Infants admitted to NICU directly or via NBN would have vital signs monitored as per NICU nursing protocol until discharge 13. Documentation of Length of Stay in NBN or NICU will collected 14. Documentation of intensity of care, type of support, maximum FiO2 required and duration of respiratory support in NICU will be collected.

ELIGIBILITY:
Inclusion Criteria:

* Obstetrical patients delivering at Weiler Hospital.
* Any woman not in labor, who is undergoing scheduled caesarean deliveries at term (37 - 42 completed weeks of gestation),

Exclusion Criteria:

* Women with prior rupture of membranes
* Women receiving magnesium sulfate
* Women with known illegal drug history
* fetus with known congenital anomalies or if meconium stained fluid is present.
* mother with maternal fever, chorioamnionitis
* babies experiencing fetal distress e.g. abnormal fetal heart tracing,
* non vigorous newborn at birth (defined as per NRP guidelines as infant with apnea/gasping, heart rate <100/min, poor tone).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 500 (Actual)
Dates: Start 2015-12; Primary Completion 2018-12-02 (Actual); Study Completion 2018-12-18 (Actual)

PRIMARY OUTCOMES:
Administration of positive pressure ventilation and/or oxygen in prone vs supine groups | 30 minutes
  any administration of positive pressure ventilation and /or oxygen

SECONDARY OUTCOMES:
Differences in pulse oximetry recordings between prone and supine groups | 5 minutes
  Investigators will record saturations in % at 1 min, 2 min, 3 min, 4 min, 5 min intervals and compare between the groups.
Differences in heart rate between prone and supine groups | 5 minutes
  Investigators will record heart rate (beats/minute) at 1 min, 2 min, 3 min, 4 min, 5 min time points
Differences in respiratory rate between prone and supine groups | 5 minutes
  Investigators will record respiratory rate (beats/minute) at 1 min, 2 min, 3 min, 4 min, 5 min time points
Differences in neonatal intensive care admission rates between prone and supine groups | 30 minutes
  Neonatal resuscitation team leader makes the decision regarding neonatal intensive care admission need as per Weiler Hospital/Montefiore guidelines; rates will be compared between the two groups.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Havranek, MD, Principal Investigator — Albert Einstein University/Montefiore Medical Center
Locations (1):
- Weiler Hospital, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: No